CLINICAL TRIAL: NCT00597272
Title: Pilot Trials With a KLH Conjugated Bivalent GangliosideVaccine Mixed With Immunological Adjuvants QS-DG or OPT-821in Patients With Disease Free AJCC Stage III or IV
Brief Title: Determine Toxicity and Antibody Responses With a KLH Conjugated Bivalent Vaccine Containing GD2 Lactone, GD3 Lactone With Immunological Adjuvant QS-DG or OPT-821 in Patients With Disease Free AJCC Stage III or IV Cutaneous Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-086
Record Dates: First submitted 2008-01-08; First posted 2008-01-18 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Melanoma
Keywords: melanoma; resected local; systemic metastasis
MeSH Terms: conditions — Melanoma

ARMS (1):
- 1 (Experimental): Vaccine- KLH conjugates with GD2L and GD3L
  Interventions: Biological: KLH conjugates with GD2L and GD3L

INTERVENTIONS:
Biological: KLH conjugates with GD2L and GD3L — 6 vaccinations (on weeks 1, 2, 3, 8, 20 and 32) which will contain the same KLH conjugates with GD2L and GD3L. All vaccines contain KLH conjugates containing 30mcg of GD2L and 30mcg of GD3L and QS-DG or OPT-821. The initial 8 patients will receive the same QS-DG or OPT-821 vaccine dose in all of their vaccines. This dose will be 50 mcg for the first patient, 75 mcg for the second patient and 100 mcg for the third through eighth patients. In all subsequent patients the 1st, 4th and 5th vaccinations will include 150 mcg of OPT-821. The 2nd and 3rd vaccinations will contain 100 mcg of OPT-821 and the 6th vaccination will contain 200 mcg of OPT-821.

SUMMARY:
Vaccines contain substances that help us make antibodies. Different antibodies help protect us against a variety of harmful things. GD2 and GD3 gangliosides are substances found on the surface of most melanoma cells. They are also occasionally found on some normal cells. Large quantities of antibodies called monoclonal antibodies have been prepared in the laboratory against GD2 and GD3 and given to patients with metastatic melanoma. In about 10% of cases this has resulted in clinically relevant regression of melanomas. These monoclonal antibodies are not currently available or used in the clinic but studies in the laboratory indicate that vaccines against GD2 and GD3 can be as effective as monoclonal antibodies.

In this trial we wish to raise the level of antibodies in your blood against GD2 and GD3. We will vaccinate you with the modified forms of GD2 called GD2 lactone and GD3 called GD3 lactone (GD3L), all attached to the antibody booster KLH, and mixed with the immune booster (immunologic adjuvant) QS-DG. While over a thousand patients have received vaccines with QS-21, the QS-DG used here is synthesized for the first time at MSKCC and is referred to as QS-DG rather than QS-21 which is purified from tree bark. QS-21 and QS-DG are, to the best of our knowledge chemically identical. It is unknown if using this bivalent vaccine will raise the level of antibodies in your blood to either ganglioside. It is unknown if raising the level of antibodies in your blood will lower your risk of relapse. This study will check your blood for production of antibodies, and check you for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 with AJCC stage III or IV melanoma two weeks to one year after becoming clinically free of disease will be eligible.
* For all patients' pathology slides must be reviewed by the Memorial Hospital Department of Pathology to confirm diagnosis of cutaneous melanoma.
* All patients must have a Karnofsky performance status of ≥80.
* Patients may have received previous radiation, chemotherapy or systemic immunotherapy (completed at least 4 weeks prior to vaccination).
* A CBC must be performed within 2 weeks prior to vaccination with the WBC > or equal to 3.0 cells/mm3, Platelets >100,000/mm3,
* A screening profile must be performed within 2 weeks prior to vaccination with the total bilirubin ≤ 2.0, and other LFTs within normal limits for patient's age.
* Chest, abdomen and pelvic CT or MRI must be performed within 4 weeks of the initiation of treatment showing no evidence of disease.
* Women of child bearing potential and sexually active males must be counseled to use an accepted and effective method of contraception (including abstinence) while on treatment.

Exclusion Criteria:

* Patients previously treated with KLH or ganglioside containing vaccines, or monoclonal antibodies against gangliosides are not eligible.
* Women must not be pregnant (negative βHCG within 2 weeks of vaccination if of childbearing potential).
* Patients with other active cancers within the past 2 years, (excluding basal cell, squamous carcinomas of the skin or cervical carcinoma-in-situ) are not eligible.
* Any medical condition which might make it difficult for the patient to complete the full course of treatments or to respond immunologically to them is grounds for exclusion, at the discretion of the Principal Investigator.
* Patients requiring anti-inflammatory medications such a steroids, NSAIDS or full dose aspirin are not eligible.
* There must be no evidence of metastatic disease at the time of the first vaccine. However, patients who develop new metastases during treatment may continue on treatment as long as no systemic treatment is indicated and any local treatment such as surgical resection or radiation would not cause a delay in vaccination or two weeks or more.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1A: Cohort 1A: 50mcg OPT-821 weeks 1, 2, 3, 8, 20, 32
- Cohort 1B: Cohort 1B: 75mcg OPT-821 weeks 1, 2, 3, 8, 20, 32
- Cohort 1C: Cohort 1C: 100mcg OPT-821 weeks 1, 2, 3, 8, 20, 32
- Cohort 2A: Cohort 2A: 50mcg QS-DG weeks 1, 2, 3, 8, 20, 32
- Cohort 2B: Cohort 2B: 75mcg QS-DG weeks 1, 2, 3, 8, 20 ,32
- Cohort 2C: Cohort 2C: 100mcg QS-DG weeks 1, 2, 3, 8, 20 ,32
- Cohort 3: Cohort 3: 150mcg OPT-821 for first 5 vaccines with a 50 mcg increase in dose for the final vaccine.
Period: Overall Study
Arm/Group | Cohort 1A | Cohort 1B | Cohort 1C | Cohort 2A | Cohort 2B | Cohort 2C | Cohort 3
Started | 1 | 1 | 10 | 1 | 1 | 10 | 10
Completed | 1 | 1 | 10 | 1 | 1 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A | Cohort 1B | Cohort 1C | Cohort 2A | Cohort 2B | Cohort 2C | Cohort 3 | Total
Number analyzed (Participants) | 1 | 1 | 10 | 1 | 1 | 10 | 10 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 8 | 1 | 1 | 8 | 8 | 27
  >=65 years | 1 | 0 | 2 | 0 | 0 | 2 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 4 | 0 | 0 | 5 | 1 | 11
  Male | 0 | 1 | 6 | 1 | 1 | 5 | 9 | 23
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 10 | 1 | 1 | 10 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Toxicity will be graded in accordance with Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Cohort 1A | Cohort 1B | Cohort 1C | Cohort 2A | Cohort 2B | Cohort 2C | Cohort 3
Number analyzed (Participants) | 1 | 1 | 10 | 1 | 1 | 10 | 10
participants | 1 | 1 | 6 | 1 | 1 | 7 | 10

ADVERSE EVENTS:
Arm/Group | Cohort 1A | Cohort 1B | Cohort 1C | Cohort 2A | Cohort 2B | Cohort 2C | Cohort 3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/10 | 0/1 | 0/1 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 6/10 | 1/1 | 1/1 | 7/10 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A (N=1) | Cohort 1B (N=1) | Cohort 1C (N=10) | Cohort 2A (N=1) | Cohort 2B (N=1) | Cohort 2C (N=10) | Cohort 3 (N=10)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 1 (5) | 1 (1) | 1 (4) | 2 (2) | 1 (1)
Injection site reaction (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 9 (32)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inf unknown ANC-Pneumonia(lung) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection w/ Gr 3/4 neut, Dental-tooth (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes